CLINICAL TRIAL: NCT02197507
Title: Evaluation of Grip Strength With Digitized Sensor in Adults With Rheumatoid Arthritis
Brief Title: Digitized Grip Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9385
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RA patients (Experimental)
  Interventions: Device: Digitized sensor

INTERVENTIONS:
Device: Digitized sensor — Measure of grip strength of the dominant hand

SUMMARY:
Rheumatoid arthritis (RA) is the most common chronic inflammatory arthritis in adults. Monitoring of disease activity is based on Disease Activity Score 28 (DAS 28). There are also validated questionnaires for self-assessment of the disease by the patient. Grip strength measured using a digitized sensor used by the patient could be an additional tool to the remote monitoring of patients with RA.

Main Objective : To evaluate the correlation between the measurement of grip strength in the dominant hand measured by a digital sensor and activity of RA assessed by DAS 28

Secondary objective : Evaluate the correlation between grip strength of the dominant hand and :

* scores of fatigue and pain (VAS and FACIT)
* the self-assessment scores known in RA : functional index Health Assessment Questionnaire (HAQ) and scores of activity RAPID3 and RADAI5.

It is a cross-sectional study involving 150 patients followed in our department for RA. Grip strength of the dominant hand will be measured by a digitalized sensor during a single visit integrating into the routine monitoring of patients.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis whatever its activity
* Above 18 years old patients

Exclusion Criteria:

* Other condition that may affect the level of fatigue and / or grip strength
* Insufficient level of understanding to perform the measurement and self-report questionnaires

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
grip strength | visit 1
  Evaluate the correlation between the measurement of grip strength in the dominant hand measured by a digital sensor and activity of RA assessed by DAS 28

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France